CLINICAL TRIAL: NCT03164551
Title: A Phase IV, Single-blinded, Prospective, Randomized, Controlled, Multi-center Study to Compare the Clinical Outcomes of Genea Embryo Review Instrument Plus (GERI+) Time Lapse System With a Conventional Embryo Culture and Assessment System
Brief Title: TICON-Day 3, Time Lapse Versus Conventional Method in Day 3 Embryo Culture and Assessment
Acronym: TICON
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Participant enrollment has remained significantly behind plan despite increased site enrollment activity.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS200497_0006
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Infertility
Keywords: GERI+; TICON; EEVA; Embryo culture; In Vitro Fertilization; Intracytoplasmic Sperm Injection
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GERI+ Incubator (Active Comparator)
  Interventions: Device: GERI+ incubator
- Conventional incubator (Other)
  Interventions: Device: Conventional incubator

INTERVENTIONS:
Device: GERI+ incubator — The embryo culture of consented participants were carried out in GERI+ incubator for both bright-field and dark-field time lapse monitoring until Day 3 of embryo culture. On Day 3, all embryos were reviewed firstly by GERI Assess software, using bright-field imaging. Finally the embryo(s) with the highest EEVA grade are transferred were followed up until the achievement of implantation and confirmation of pregnancy.
  Arms: GERI+ Incubator
Device: Conventional incubator — The embryo culture of consented participants were carried out in conventional incubator for culture until Day 3 of embryo culture. On Day 3 of embryo culture, all embryos are assessed using a bench-top microscope. The embryo(s) with optimal cell stage and grade were transferred and were followed up until the achievement of implantation and confirmation of pregnancy.
  Arms: Conventional incubator

SUMMARY:
The main purpose of the study was to evaluate the overall clinical value of GERI+ as an integrated embryo culture and assessment system, providing an undisturbed culture environment, continuous monitoring of embryo development and automated scoring using a predictive algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Couples with less than or equal to (<= ) two failed fresh In Vitro Fertilization/Intracytoplasmic Sperm Injection (IVF/ICSI) embryo transfer cycles
* Age greater than or equal to (>=) 18 and <= 40 years
* Body mass index (BMI): 18-30 kilogram per meter square (kg/m2)
* Normal uterine cavity under ultrasound
* Participant and her husband/partner must have read and signed the Informed Consent form (ICF)
* At least four normally fertilized oocytes (2Pronuclear stage (PN)) in the current cycle

Exclusion Criteria:

* Male with non-ejaculated sperm
* Participants with abnormal, undiagnosed gynecological bleeding or with genitourinary malformations
* Participants with any contraindication to Controlled Ovarian Stimulation (COS) for Assisted Reproductive Technologies (ART) or to gonadotropins
* Planned "freeze all" cycle (oocytes or embryos)
* Planned preimplantation genetic screening (PGS) or Pre-implantation genetic diagnosis (PGD) cycle
* Concurrent participation in another clinical study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 408 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (17):
- Canada (2):
  - Cambrian Wellness Centre, Calgary
  - Regional Fertility Program, Calgary
- Denmark (2):
  - Skive Fertility clinic, Skive
  - Fertility Clinic Skive Regional Hospital, Skive
- Hopital Antoine Beclere, Clamart, France
- Italy (4):
  - Krankenhaus Bruneck, Bruneck (BZ)
  - Demetra S.R.L, Florence
  - Futura Diagnostica medica PMA SRL, Florence
  - USL Toscana Nordovest, Viareggio
- Norway (3):
  - Oslo University Hospital, Oslo
  - Sykehuset Telemark HF Fertilitetsavdeliningen Sor, Skien
  - St. Olavs Hospital Hf, Universitetssykehuset i Trondheim, Trodheim
- Centro Hospitalar e Universitario de Coimbra, Coimbra, Portugal
- Spain (4):
  - Hospital de Cruces, Barakaldo
  - Nephrology Service Fundacion Puigvert, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hosp Univ de Canarias, Santa Cruz de Tenerife

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200497_0006
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- GERI+ Incubator: The embryo culture of consented participants carried out in Genea Embryo Review Instrument Plus (GERI+) incubator for both bright-field and dark-field time lapse monitoring until Day 3 of embryo culture. On Day 3, all embryos were reviewed firstly by GERI Assess software, using bright-field imaging. Finally the embryo(s) with the highest EEVA grade were transferred and were followed up until the achievement of implantation and confirmation of pregnancy.
- Conventional Incubator: The embryo culture of consented participants were carried out in conventional incubator for culture until Day 3 of embryo culture. On Day 3 of embryo culture, all embryos were assessed using a bench-top microscope. The embryo(s) with optimal cell stage and grade were transferred and were followed up until the achievement of implantation and confirmation of pregnancy.
Period: Overall Study
Arm/Group | GERI+ Incubator | Conventional Incubator
Started | 200 | 208
Completed | 171 | 192
Not Completed | 29 | 16
Not completed — Imaging discontinued prior completion | 8 | 0
Not completed — Participant was non-compliant | 1 | 0
Not completed — Cancellation of Fresh Embryo Transfer | 12 | 14
Not completed — Other | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GERI+ Incubator | Conventional Incubator | Total
Number analyzed (Participants) | 200 | 208 | 408
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.27 (4.076) | 33.23 (3.996) | 33.25 (4.030)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 208 | 408
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy Rate With Positive Fetal Heart Beat (FHB)
Description: Clinical Pregnancy was defined as the pregnancy diagnosed by ultrasonographic or clinical documentation of at least one fetus with heart beat in gestational week 6 to 8. Clinical pregnancy rate with positive FHB was measured as the number of participants with FHB positive clinical pregnancy divided by number of participants with embryo transfer (ET) multiplied by 100. Here, data used for analysis was based on Merck Global Medical Affairs (GMA) interpretation.
Time Frame: Gestation Weeks 6 to 8
Population: Full analysis (FA) dataset included all randomized participants.
Measure: Number; unit: Percentage of pregnancy per ET
Arm/Group | GERI+ Incubator | Conventional Incubator
Number analyzed (Participants) | 200 | 208
Percentage of pregnancy per ET | 39.4 | 38.9

2. Secondary Outcome: Utilizable Embryos Rate
Description: Utilizable embryos rate is defined as the number of transferred and cryopreserved embryos divided by the number embryos stage zygotes per participant multiply by 100. Here, data used for analysis was based on Merck GMA interpretation.
Time Frame: Day 3 of embryo culture
Population: FA dataset included all randomized participants. Here, "Number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of embryos
Arm/Group | GERI+ Incubator | Conventional Incubator
Number analyzed (Participants) | 198 | 208
Percentage of embryos | 50.72 (23.379) | 50.11 (24.183)

3. Secondary Outcome: Good Quality Embryos Rate
Description: Good Quality Embryos is defined embryos with 7 or more blastomeres, less than (<) 25 % fragmentation, size and symmetry of blastomeres appropriate to the cell number, and no evidence of multinucleation, based on the morphology on Day 3 of embryo culture. Good quality embryos rate was defined as the number of good quality embryos divided by the number of embryos per participant multiplied by 100. Here, data used for analysis was based on Merck GMA interpretation.
Time Frame: Day 3 of embryo culture
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of Good Quality Embryos
Arm/Group | GERI+ Incubator | Conventional Incubator
Number analyzed (Participants) | 198 | 208
Percentage of Good Quality Embryos | 34.85 (25.999) | 37.68 (29.115)

4. Secondary Outcome: Non-viable Embryos Rate
Description: Non-viable Embryos is defined as the embryos in which development has been arrested for at least 24 hour or in which all the cells have degenerated or lysed. Non-viable embryos rate was defined as the number of non-viable embryos divided by the number of embryos per participant multiplied by 100. Here, data used for analysis was based on Merck GMA interpretation.
Time Frame: Days 1 to 3 of embryo culture
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of Non-viable Embryos
Arm/Group | GERI+ Incubator | Conventional Incubator
Number analyzed (Participants) | 198 | 208
Percentage of Non-viable Embryos | 29.64 (27.932) | 30.67 (29.001)

5. Secondary Outcome: Implantation Rate (IR) With Positive Fetal Heart Beat
Description: A successful implantation is defined as the presence of one gestational sac with fetal heart beat (FHB) under ultrasonography at gestational weeks 6-8. Implantation rate (IR) was defined as the number of intrauterine gestational sacs with positive FHB under ultrasound scans at gestational weeks 6-8 divided by the total number of embryos transferred (ET) multiplied by 100. Here, data used for analysis was based on Merck GMA interpretation.
Time Frame: Gestational Weeks 6 to 8
Population: FA dataset included all randomized participants.
Measure: Number; unit: Percentage of gestational sacs per ET
Arm/Group | GERI+ Incubator | Conventional Incubator
Number analyzed (Participants) | 200 | 208
Percentage of gestational sacs per ET | 31.2 | 32.5

6. Secondary Outcome: Biochemical Pregnancy Rate
Description: Biochemical Pregnancy defined as a pregnancy diagnosed only by the detection of Human Chorionic Gonadotropin (hCG) in serum or urine and that does not develop into a clinical pregnancy. Biochemical pregnancy rate was defined as the number of participants with biochemical pregnancy divided by the number of participants with embryo transfer (ET) multiplied by 100. Here, data used for analysis was based on Merck GMA interpretation.
Time Frame: From Day 12 of Gestational up to Week 8
Population: FA dataset included all randomized participants.
Measure: Number; unit: Percentage of Pregnancy per ET
Arm/Group | GERI+ Incubator | Conventional Incubator
Number analyzed (Participants) | 200 | 208
Percentage of Pregnancy per ET | 7.2 | 4.7

7. Secondary Outcome: Ongoing Pregnancy Rate
Description: Ongoing pregnancy is defined as the presence of viable fetuses identified by ultrasonography at gestational weeks 10-12. Ongoing pregnancy rate is defined as the number of participants with ongoing pregnancy divided by the number of participants with embryo transfer (ET) multiplied by 100. Here, data used for analysis was based on Merck GMA interpretation.
Time Frame: Gestational Weeks 10 to 12
Population: FA dataset included all randomized participants.
Measure: Number; unit: Percentage of Pregnancy per ET
Arm/Group | GERI+ Incubator | Conventional Incubator
Number analyzed (Participants) | 200 | 208
Percentage of Pregnancy per ET | 35.0 | 36.3

8. Secondary Outcome: Multiple Pregnancy Rate
Description: Multiple pregnancy is defined as a pregnancy with more than one fetus. It is identified by ultrasonography at gestational weeks 10-12. Multiple pregnancy rate was defined as the number of participants with multiple pregnancy divided by the number of participants with ongoing pregnancy multiplied by 100. Here, data used for analysis was based on Merck GMA interpretation.
Time Frame: Gestational Weeks 10 to 12
Population: FA dataset included all randomized participants.
Measure: Number; unit: Percentage of Multiple Pregnancy
Arm/Group | GERI+ Incubator | Conventional Incubator
Number analyzed (Participants) | 200 | 208
Percentage of Multiple Pregnancy | 1.6 | 11.4

9. Secondary Outcome: Ectopic Pregnancy Rate
Description: Ectopic pregnancy is defined as a pregnancy in which implantation takes place outside the uterine cavity. It is identified by ultrasonography at weeks 6-8. Ectopic Pregnancy Rate was defined as the number of participants with ectopic pregnancy divided by the number of participants with embryo transfer (ET) multiplied by 100. Here, data used for analysis was based on Merck GMA interpretation.
Time Frame: Gestational Weeks 6 to 8
Population: FA dataset included all randomized participants.
Measure: Number; unit: Percentage of Pregnancy per ET
Arm/Group | GERI+ Incubator | Conventional Incubator
Number analyzed (Participants) | 200 | 208
Percentage of Pregnancy per ET | 1.1 | 0.5

10. Secondary Outcome: Spontaneous Miscarriage Rate
Description: Spontaneous miscarriage (SM) is the spontaneous loss of a clinical pregnancy before 20 completed weeks of gestational age (18 weeks after fertilization). In this study, the spontaneous miscarriage was tracked up to 10-12 weeks of gestational age. Spontaneous miscarriage rate was defined as the number of participants with spontaneous miscarriage divided by the number of participants with clinical pregnancy multiplied by 100. Here, data used for analysis was based on Merck GMA interpretation.
Time Frame: Gestational Weeks 10 to 12
Population: FA dataset included all randomized participants.
Measure: Number; unit: Percentage of miscarriages
Arm/Group | GERI+ Incubator | Conventional Incubator
Number analyzed (Participants) | 200 | 208
Percentage of miscarriages | 9.3 | 10.1

ADVERSE EVENTS:
Time Frame: Not Applicable (NA)
Description: This is a fertility device technology study and this study was not designed to monitor all-cause mortality, serious, and other (not Including serious) adverse events. Therefore, all-cause mortality, serious, and other (not Including serious) adverse events data could not be reported.
Arm/Group | GERI+ Incubator | Conventional Incubator
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT03164551/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT03164551/SAP_001.pdf